CLINICAL TRIAL: NCT05549609
Title: A Multi-centre, Randomised, Single-blind Phase I/IIa Study to Evaluate the Safety, Tolerability and Efficacy of a Single Topical Dose of Allogeneic Integrin α10β1-selected Mesenchymal Stem Cells (XSTEM-VLU) in Patients With Difficult-to-heal Venous Leg Ulcers
Brief Title: A Study of XSTEM-VLU in Patients With Difficult-to-heal Venous Leg Ulcers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xintela AB (Industry)
Collaborators: Vinnova (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XIN-XSTEM-201
Record Dates: First submitted 2022-09-06; First posted 2022-09-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XSTEM-VLU (Experimental): Single topical dose of XSTEM-VLU
  Interventions: Biological: XSTEM-VLU
- Vehicle (Placebo Comparator): Single topical dose of CryoStor CS10
  Interventions: Other: Vehicle

INTERVENTIONS:
Biological: XSTEM-VLU — XSTEM-VLU is an allogeneic, adipose tissue-derived, integrin alpha10beta1-selected and expanded mesenchymal stem cell (MSC) product for the treatment of venous leg ulcers.
  Arms: XSTEM-VLU
Other: Vehicle — CryoStor CS10 cryomedium
  Arms: Vehicle

SUMMARY:
The aim of the study is to assess safety, tolerability and preliminary efficacy of XSTEM-VLU when administered as a single topical dose to patients with difficult-to-heal venous leg ulcers. The study is randomised and the patients will receive either XSTEM-VLU or vehicle as add on to standard wound care.

The patients will be followed weekly for 10 weeks after treatment. At 4 months after treatment, the patients will return to the clinic for an end-of-study visit.

ELIGIBILITY:
Major Inclusion Criteria:

* Written informed consent for participation in the study
* Male or female patient aged ≥18 years
* BMI ≥18.5 and ≥40.0 kg/m2
* Lower leg wound due to venous insufficiency
* Target wound has failed to heal despite standard wound care for a minimum of 6 weeks
* A surface area of the target wound of ≥2 and ≤40 cm2

Major Exclusion Criteria:

* Signs or symptoms of clinically significant ongoing infection i the target wound requiring anti-microbial treatment
* History of autoimmune disease, such as but not limited to systemic lupus erythematosus, Addison's disease, Crohn's disease and type I diabetes mellitus
* B-HbA1C value ≥52 mmol/mol
* Plaque psoriasis or any other skin disease that could interfere with the outcome of the study
* Arterial insufficiency
* History of any malignancy within the past 5 years
* Target wound diagnosed as a malignant wound, neuropathic wound, pressure wound or osteomyelitis
* Patients who are immunocompromised due to disease or for other reasons such as the use of systemic immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AEs) | From study start to 4 months after dosing
  Frequency, seriousness and intensity of AEs assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Safety and tolerability: Local tolerability | From study start to 4 months after dosing
  Local tolerability evaluated by direct inspection by need for debridement (Yes/No) and clinical signs of wound infection (Yes/No)
Safety and tolerability: Number of participants with abnormal 12-lead electrocardiogram (ECG) | From study start to 4 months after dosing
  Abnormal findings assessed by the Investigator as clinically significant will be reported as AEs.
Safety and tolerability: Number of participants with abnormal vital signs | From study start to 4 months after dosing
  Vital signs include blood pressure, pulse and body temperature. Abnormal findings assessed by the Investigator as clinically significant will be reported as AEs.
Safety and tolerability: Number of participants with abnormal laboratory test results | From study start to 4 months after dosing
  Laboratory tests include clinical chemistry, haematology and coagulation parameters. Abnormal values assessed by the Investigator as clinically significant will be reported as AEs.
Safety and tolerability: Number of participants with abnormal physical examination findings | From study start to 4 months after dosing
  Abnormal findings assessed by the Investigator as clinically significant will be reported as AEs.

SECONDARY OUTCOMES:
Preliminary efficacy: Wound area reduction (absolute and percentage) compared to baseline | From study start to 4 months after dosing
Preliminary efficacy: Proportion of patients with re-epithelialization of >=95% and >=50% of the wound area measured at baseline | From study start to 4 months after dosing
Preliminary efficacy: Time to re-epithelialization of >=95% and >=50% of the wound area measured at baseline | From study start to 4 months after dosing
Preliminary efficacy: Pain for target wound and the affected leg using Visual Analogue Scale (VAS) | From study start to 4 months after dosing
  The VAS consists of a 100 mm line from no pain (0 mm) to worst possible pain (100 mm).
Preliminary efficacy: Scar formation assessed by the Patient and Observer Scar Assessment Scale (POSAS) | At week 10 and at 4 months after dosing
  The POSAS is divided into two scales (for patient and for observer), each with six items scored numerically (1 -10). The lowest score "1" corresponds to normal skin.

CONTACTS AND LOCATIONS:
Overall Officials: Folke Sjöberg, Principal Investigator — Burn Centre, Linkoping University Hospital, Linkoping, Sweden
Locations (4):
- Sweden (4):
  - Clinical Trial Center (CTC), Gothenburg
  - Burn Centre, Linköping University Hospital, Linköping
  - Clinical Research Unit, Lund
  - Clinical Trial Consultants (CTC) Karolinska, Stockholm

IPD SHARING:
Plan to Share IPD: No